CLINICAL TRIAL: NCT06680687
Title: A Non-randomized Prospective Cohort Study to Improve Follow-up Adherence, Survivorship Knowledge and Late Effects Documentation at a Childhood Cancer Clinic in Western Kenya: A Study Protocol
Brief Title: Survivorship Intervention Program in Western Kenya: Study Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moi University (Other)
Collaborators: Princess Maxima Center for Pediatric Oncology (Other); Amsterdam UMC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 0004807
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Cancer; Survivorship
Keywords: Aftercare; Health Education; Patient Compliance; Surveillance
MeSH Terms: conditions — Neoplasms; Health Education; Patient Compliance | interventions — Videotape Recording; Metabolism

STUDY DESIGN:
Intervention Model Description: A caregiver control group of 50 participants receiving usual care will be recruited and sequentially, 50 caregivers will be included in the intervention group. Because follow-up adherence is also time-dependent (the risk of non-adherence increases with time), the investigators reasoned that the Educational Program should be delivered before completion of treatment, to prevent survivors getting lost to follow-up before receiving the intervention.
  Healthcare provider training will be provided to at least 75 percent of the healthcare providers that match the inclusion criteria and timing of the training will be determined by availability. The Follow-Up Form will be used to document late effects in all survivors that attend the outpatient clinic, regardless enrollment in the Educational Program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Usual Care" (No Intervention): Participants receiving "Usual Care" group (A), will be recruited during the last two months of treatment (T-2). At the end of treatment (T0), participants will complete a knowledge questionnaire and will be followed for another 24 months. At six months after treatment completion (T6), a final follow-up knowledge assessment will be conducted. Participants will be enrolled into group A until the intended sample size of 50 participants is reached. Investigators estimated to have reached this number within four to six months based on recent survival rates.
- "Educational Intervention" (Experimental): A similar procedure will apply to the "Educational Intervention" group (B). Participants will complete a knowledge assessment before receiving an educational intervention between T-2 and T0. To evaluate early and late knowledge uptake, participants will complete a post-education knowledge assessment at T0 and a follow-up knowledge assessment at T6. Follow-up adherence will be evaluated at every three months for the first year and at every six months during the second year after treatment completion for both groups. Implementation measures will be captured starting at T3 until T24, together with a satisfaction questionnaire that will be administered at T6.
  Interventions: Behavioral: Educational Program (video, information booklet, Survivorship Card)
- "Follow-Up Forms implementation" (Other): Healthcare provider training on survivorship will start at the same timepoint as recruitment of the "Educational Intervention" group (A) at T-2.
  Follow-Up Forms will be introduced at the outpatient clinic once an estimated 30 healthcare providers have done the training (anticipated at T0). Healthcare providers will fill in a knowledge assessment directly pre- and post-training (T-2) and at six months post-training (T4).
  Documentation of late effect symptoms will be monitored for twelve months, starting at T0. Implementation measures will be collected weekly starting from T0 and healthcare providers will be assigned to a satisfaction questionnaire at T6.
  Interventions: Behavioral: Follow-Up Program (form and healthcare provider training)

INTERVENTIONS:
Behavioral: Educational Program (video, information booklet, Survivorship Card) — Caregivers will be invited to attend an educational group session. Each session will be organized weekly to monthly. A maximum of ten caregivers can be present at a session.
  First a video will be displayed in which healthcare providers explain medical aspects of survivorship. Caregivers of survivors and young adult survivors discuss experiences after completing cancer treatment in the video.
  Secondly, the present healthcare provider will hand over an information booklet 'Life after childhood cancer' to the caregivers. The booklet covers similar topics as presented in the video.
  Lastly, a Survivorship Card will be shared with the caregivers. The card contains a record of the patient's cancer and treatment history and the expected follow-up appointment schedule. The survivor and family take one card home and a duplicate copy of the card remains in the medical file.
  Arms: "Educational Intervention"
Behavioral: Follow-Up Program (form and healthcare provider training) — Healthcare providers will attend a training session of approximately 90 minutes, in which investigators will discuss the same topics as covered in the educational group session supported by PowerPoint slides.
  A Follow-Up Form will be introduced to be used by healthcare providers in the outpatient follow-up clinic. The form will include questions referring to symptoms specific for certain late effects. Specific questions will be included per subcategory: hematological malignancies, solid tumors or central nervous system (CNS) tumors.
  Arms: "Follow-Up Forms implementation"

SUMMARY:
In this study protocol, the investigators described a survivorship intervention program that will be performed at a referral hospital in Western Kenya. This will be a non-randomized prospective cohort study with a sequential hybrid effectiveness - implementation design. The study comprises of an educational component for caregivers of childhood cancer survivors and a follow-up component targeting healthcare providers with survivorship training and implementation of a late effects documentation tool.

Through these interventions the investigators aim to:

1. increase follow-up adherence of childhood cancer survivors;
2. increase caregivers' and healthcare providers' knowledge about childhood cancer diagnoses, treatment and the corresponding late effects risks;
3. document late effects at a childhood cancer outpatient clinic;
4. evaluate program implementation and satisfaction among recipients and providers.

DETAILED DESCRIPTION:
This non-randomized prospective cohort study will be performed at a referral hospital in Western Kenya. Hundred caregivers of children diagnosed with cancer, who will complete treatment within two months, will be enrolled and followed for 24 months after completion of treatment. A caregiver control group receiving usual care will be recruited and sequentially, caregivers will be included in an intervention group to attend an educational group session and receive educational materials (video, booklet and Survivorship Card). Primary study outcome will be survivors' follow-up adherence. Survivors will be considered lost to follow-up after missing a scheduled appointment and subsequently do not revisit the clinic for more than six months. Mixed models regression analyses will be performed to determine intervention effects on follow-up adherence and secondly on caregiver survivorship knowledge uptake. Additionally, healthcare providers will be trained on follow-up care, whereafter a form will be introduced at the outpatient clinic to document late effects in pediatric survivors attending the clinic for the period of a year. Secondary outcomes will be late effects prevalence as documented in the Follow-Up Form and healthcare provider survivorship knowledge uptake. Implementation measures (reach, potential effectiveness, adoption, satisfaction and maintenance) will be evaluated for both programs.

ELIGIBILITY:
Inclusion criteria:

* Caregivers of children diagnosed with cancer (primary or secondary malignancy) below fifteen years old.
* Children will soon be finalizing childhood cancer treatment (enrolled during the last 2 months of treatment).
* Healthcare providers (the pediatric oncology workforce comprises of an estimated 30 staff members) working in the Pediatric Oncology department at MTRH will be recruited.
* Any cadre involved in patient care or patient education (e.g. pediatric oncologists, fellows, registrars, medical officers, clinical officers, nurses, patient navigators, child life specialists) will be allowed to participate.

Exclusion criteria:

* Childhood cancer patients should have no treatment failure (abandonment, relapsed disease, progressive disease).
* Caregivers of children with a relapsed malignancy in remission will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of non-adherent study participants | 24 months: at 3, 6, 9, 12, 18 and 24 months.
  When survivors do not appear at a scheduled visit within four weeks before or after the scheduled date.
Percentage of participants lost to follow-up | 24 months: at 3, 6, 9, 12, 18 and 24 months.
  When survivors miss a scheduled appointment and do not revisit the follow-up clinic after a missed appointment for more than six months.
Reasons for non-adherence (questionnaire) | 24 months: at 3, 6, 9, 12, 18 and 24 months.
  Reasons for non-adherence (death, relapse, other logistic issues) will be explored through a phone call.
Intentions to revisit the follow-up clinic (questionnaire) | 24 months: at 3, 6, 9, 12, 18 and 24 months.
  Intentions to revisit the follow-up clinic (yes/no, what can hospital do to support participant in adhering to follow-up visit) will be explored through a phone call.

SECONDARY OUTCOMES:
Caregiver knowledge (questionnaire) | Two months prior to survivor's treatment completion, assessed up to six months after completion of treatment
  Caregivers' knowledge about disease history, treatment exposure, associations between treatment and late effects, follow-up care, late effects risk and risk perception.
  Levels of knowledge (number of accurate/inaccurate/unknown responses), and knowledge uptake (changes in number of accurate responses) progression will be followed over time.
Healthcare provider knowledge (questionnaire) | From start healthcare provider training up to six months after the completion of the training session
  Caregivers' and healthcare providers' knowledge about disease history, treatment exposure, associations between treatment and late effects, follow-up care, late effects risk and risk perception according
  Levels of knowledge (number of accurate/inaccurate/unknown responses), and knowledge uptake (changes in number of accurate responses) progression will be followed over time.
Follow-Up Form documented late effects prevalence | 12 months: weekly.
  The prevalence of late effects will be described as the percentage of individual survivors visiting the outpatient clinic for the duration of one year that reported a symptom (yes/no) as documented in the follow-up forms.
  Late effects are categorized into physical outcomes (e.g. relapsed disease, heart failure), physical aspects of quality of life (e.g. fatigue, challenges exercising), psychosocial aspects of quality of life (e.g. anxiety, exclusion), neurocognitive aspects of quality of life (memory, educational problems) according to the International Childhood Cancer Outcome Project.
Reach caregivers (Implementation measures data collection tool) | 24 months: weekly
  Percentage eligible caregivers having received the booklet, video and Survivorship Card, characteristics of caregivers included in the study
Reach healthcare providers (Implementation measures data collection tool) | 12 months: weekly.
  Percentage eligible healthcare providers trained, Characteristics of healthcare providers included in the study
Adoption caregivers (Implementation measures data collection tool) | 24 months: at 3, 6, 9, 12, 18 and 24 months
  Percentage study participants taking the Survivorship Card to clinic appointment
Adoption healthcare providers (Implementation measures data collection tool) | 12 months: weekly.
  Percentage eligible survivors having received the follow-up form in clinic; Percentage follow-up forms completely filled by clinician; Investigations and referrals done; Actions adhering to form instructions
Caregiver satisfaction (questionnaire) | At 6 months after receiving the educational intervention
  Satisfaction questionnaire rating satisfaction on a 3-point Likert scale (highest score indicating maximum satisfaction, and lowest score indicating maximum satisfaction for inverse questions). Values can range from minimum 1 (Disagree) to maximum 3 (Agree).
Healthcare provider satisfaction (questionnaire) | At 6 months after receiving the healthcare provider training
  Satisfaction questionnaire rating satisfaction on a 5-point Likert scale (highest score indicating maximum satisfaction, and lowest score indicating maximum satisfaction for inverse questions). Values can range from minimum 1 (Strongly Disagree) to maximum 5 (Strongly Agree).
Caregiver recommendations | At 6 months after receiving the educational intervention
  Open question exploring recommendations to improve educational intervention
Healthcare provider recommendations | At 6 months after receiving the healthcare provider training
  Open question exploring recommendations to improve the Follow-Up Form

CONTACTS AND LOCATIONS:
Overall Officials: Festus Njuguna, MD, PhD, Principal Investigator — Moi University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Rift Valley, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the corresponding authors upon reasonable request after publication of all results reporting on the the Primary and Secondary Outcomes of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No end date
Access Criteria: Any reasonable request to access underlying study data

REFERENCES:
- [Derived] Lemmen J, Mageto S, Vik T, Olbara G, Kaspers G, Njuguna F. Non-randomised prospective clinical trial to improve follow-up adherence, survivorship knowledge and late effects documentation at a childhood cancer clinic in Western Kenya: a study protocol. BMJ Open. 2025 Jun 10;15(6):e096741. doi: 10.1136/bmjopen-2024-096741. PMID 40499965

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT06680687/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT06680687/ICF_001.pdf